CLINICAL TRIAL: NCT01663974
Title: Evaluation of Sub-syndromal Symptoms After Acute Depressive Episode in Bipolar Disorder
Acronym: POLARIS
Status: Terminated | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NFR-XXX-2012/1
Record Dates: First submitted 2012-08-07; First posted 2012-08-14 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Bipolar Disorder; Sub-syndromal Symptoms
Keywords: Bipolar Disorders; Sub-syndromal symptoms; Acute depressive episode; Symptomatic remission; Functioning remission
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bipolar disorder patients

SUMMARY:
The study aims to evaluate:

* the frequency of subsyndromal symptoms or disorders observed during interepisode phases in bipolar patients, particularly after a depressive episode in which these subsyndromal disorders are the most frequent
* the functional impact of these disorders, factors or symptom thresholds associated with functional remission, and factors associated with symptomatic remission over a sufficient follow-up (12 months).

DETAILED DESCRIPTION:
Evaluation of sub-syndromal symptoms after acute depressive episode in bipolar disorder

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with a diagnosis of bipolar disorder according to DSM-IV criteria currently followed up by the investigator in hospital or open-care practice and informed of his/her disease.
* For whom the previous episode was a bipolar depression assessed clinically stabilized for at least 4 weeks by the investigator.
* Able to complete the self-assessment diary weekly

Exclusion Criteria:

* Pregnant women.
* Patient included in a clinical trial on an investigational drug or having received an investigational drug in the preceding 30 days.
* Person deprived of freedom or subject to a guardianship (or ward) order or unable to undergo medical monitoring for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital/medico-psychological centre (CMP) [clinic] / private practice
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The prevalence of sub-syndromal symptoms after an acute depressive episode in Bipolar Disorder patients, as measured by scoring on YMRS and MADRS scales and MVAS-BP self-administered questionnaire. | 12 months
  The 10 items of the MADRS are scored as 0, 2, 4 and 6 (0 = no depressive symptoms; 6 = severe depressive symptoms). Total scores, ranging from 0 to 60, will be calculated by adding the values for the 10 items. The YMRS scale is composed of 11 items, scored from 0 to 4 (0 = no manic symptoms; 4 = severe manic symptoms). Total scores will be calculated by adding the scores for the 11 items. MVAS-BP questionnaire is composed of 26 visual analogue scales, each item is scored from 0 (extreme depressive pole) to 100 (extreme manic pole). Absence of symptoms is at the middle of the scale (value 50).

SECONDARY OUTCOMES:
Impact of sub-syndromal symptoms on functioning of real-life French Bipolar Disorder patients as measured by scoring on Functioning Assessment Short Test (FAST) scale. | 12 months
  Functioning Assessment Short Test (FAST) is a brief instrument designed to assess the main functioning problems experienced by psychiatric patients. The 24 items of the FAST questionnaire are scored from 0 to 3 (a score of 0 indicates that the patient does not experience any difficulties, while a score of 3 indicates that the patient experiences major difficulties). Total scores will be calculated by adding the scores for each item. Functional remission will be evaluated on the FAST scale ; functional remission will be defined as a score < 11 on the FAST questionnaire.
Number and type of factors associated with a symptomatic and functioning remission after recovery from an acute depressive bipolar episode in real-life French population. | 12 months
Description of the management patterns (such as number and drug-class of treatments, number and type of resource used) associated with the presence and absence of sub-syndromal symptoms after an acute bipolar depressive episode. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: J M AZORIN, Professor, Principal Investigator — Hopital Sainte Marguerite - MARSEILLE - FRANCE; A SOLVET, Doctor, Study Director — AstraZeneca - FRANCE
Locations (86):
- France (86):
  - Research Site, Aix-en-Provence
  - Research Site, Ajaccio
  - Research Site, Altkirch
  - Research Site, Armentières
  - Research Site, Avignon
  - Research Site, Bailleul
  - Research Site, Bohars
  - Research Site, Bordeaux
  - Research Site, Bourg-en-Bresse
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Cahors
  - Research Site, Castries
  - Research Site, Challes-les-Eaux
  - Research Site, Châteaulin
  - Research Site, Clermont-Ferrand
  - Research Site, Colmar
  - Research Site, Conty
  - Research Site, Coulommiers
  - Research Site, Créteil
  - Research Site, Crosne
  - Research Site, Dax
  - Research Site, Décines-Charpieu
  - Research Site, Digne-les-Bains
  - Research Site, Douai
  - Research Site, Durtol
  - Research Site, Dury
  - Research Site, Fains-Véel
  - Research Site, Fitz-James
  - Research Site, Grenoble
  - Research Site, Hazebrouck
  - Research Site, Héricourt
  - Research Site, Issoudun
  - Research Site, La Roche-sur-Foron
  - Research Site, La Roche-sur-Yon
  - Research Site, La Rochelle
  - Research Site, La Tronche
  - Research Site, La Varenne-Saint-Hilaire
  - Research Site, Lamballe
  - Research Site, Laval
  - Research Site, Le Mans
  - Research Site, Le Puy-en-Velay
  - Research Site, Le Vésinet
  - Research Site, Libourne
  - Research Site, Limoges
  - Research Site, Luynes
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Mayenne
  - Research Site, Metz
  - Research Site, Monaco
  - Research Site, Mont-de-Marsan
  - Research Site, Montfermeil
  - Research Site, Montmorency
  - Research Site, Montpellier
  - Research Site, Nancy
  - Research Site, Nemours
  - Research Site, Nevers
  - Research Site, Nice
  - Research Site, Noisiel
  - Research Site, Novillars
  - Research Site, Paimpol
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Reims
  - Research Site, Rouffach
  - Research Site, Rueil-Malmaison
  - Research Site, Saint-Denis
  - Research Site, Saint-Denis-lès-Bourg
  - Research Site, Saint-Dizier
  - Research Site, Saint-Égrève
  - Research Site, Saint-Nazaire
  - Research Site, Saint-Vincent-de-Tyrosse
  - Research Site, Sallanches
  - Research Site, Sevrey
  - Research Site, Soissons
  - Research Site, Sotteville-lès-Rouen
  - Research Site, Strasbourg
  - Research Site, Thuir
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Valence
  - Research Site, Vernon
  - Research Site, Versailles
  - Research Site, Vincennes

REFERENCES:
- See also: NIS-NFR-XXX-2012-1_Clinical_Study_Report_Synopsis.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=929&filename=NIS-NFR-XXX-2012-1_Clinical_Study_Report_Synopsis.pdf